CLINICAL TRIAL: NCT05190367
Title: Influence of Trauma on Pain Area and Widespreadness in Chronic Pain Patients
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Manuel Sanchez, Jorge, Principal Investigator, Hannover Medical School
Other Study IDs: 9681
Record Dates: First submitted 2021-12-10; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Chronic Pain; Trauma
MeSH Terms: conditions — Chronic Pain; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- No trauma: Patients suffering from chronic pain without traumatic life events
- Accidental trauma: Patients suffering from chronic pain who have experienced at least one accidental trauma
- Interpersonal trauma: Patients suffering from chronic pain who have experienced at least one interpersonal trauma
- PTSD: Patients suffering from chronic pain and diagnosed with PTSD

SUMMARY:
It is well known that patients suffering from chronic pain report higher levels of pain, anxiety, and depression if they have experienced a traumatic event. However, little is know about pain area and widespreadness.

In this retrospective study, we want to investigate whether pain area and widespreadness differs in chronic pain patients with and without traumatic events. To test this hypothesis we will retrospectively analyse pain drawings collected at the pain outpatient department from Hannover Medical School. Participants will be divided into four groups depending on the severity of their traumatic events: no trauma; accidental trauma; interpersonal trauma; post-traumatic stress disorder (PTSD).

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic pain visiting the pain outpatient department at Hannover Medical School.
Sampling Method: Non-Probability Sample
Enrollment: 914 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Difference in pain area | First visit of each patient at the Pain outpatient department of Hannover Medical School between 2019-02-28 and 2020-07-07
  Pain area derived from electronic pain drawings (SymptomMapper). The score ranges from 0 to 100% body area.
Difference in pain widespreadness | First visit of each patient at the Pain outpatient department of Hannover Medical School between 2019-02-28 and 2020-07-07
  Widespread pain index (WPI) derived from electronic pain drawings (SymptomMapper). The score ranges from 0 (no pain) to 19 (pain affects all possible regions).

SECONDARY OUTCOMES:
Difference in current pain | First visit of each patient at the Pain outpatient department of Hannover Medical School between 2019-02-28 and 2020-07-07
  Visual analogue scale from 0 ("no pain") to 100 ("maximal imaginable pain").
Difference in mean pain in the last four weeks | First visit of each patient at the Pain outpatient department of Hannover Medical School between 2019-02-28 and 2020-07-07
  Visual analogue scale from 0 ("no pain") to 100 ("maximal imaginable pain").
Difference in maximal pain in the last four weeks | First visit of each patient at the Pain outpatient department of Hannover Medical School between 2019-02-28 and 2020-07-07
  Visual analogue scale from 0 ("no pain") to 100 ("maximal imaginable pain").
Difference in acceptable pain | First visit of each patient at the Pain outpatient department of Hannover Medical School between 2019-02-28 and 2020-07-07
  Visual analogue scale from 0 ("no pain") to 100 ("maximal imaginable pain").
Difference in sleep impairment | First visit of each patient at the Pain outpatient department of Hannover Medical School between 2019-02-28 and 2020-07-07
  Visual analogue scale from 0 ("no impairment") to 100 ("maximal imaginable impairment").
Difference in pain-related disability | First visit of each patient at the Pain outpatient department of Hannover Medical School between 2019-02-28 and 2020-07-07
  Pain-related disability assessed via the Pain Disability Index (PDI). The score ranges from 0 (no pain-related disability) to 70 (maximal disability).
Difference in depression | First visit of each patient at the Pain outpatient department of Hannover Medical School between 2019-02-28 and 2020-07-07
  Depression assessed via the 9-item depression scale (PHQ-9) from the German version of the Patient Health Questionnaire (PHQ-D). The score ranges from 0 (no depression) to 27 (maximal depression).
Difference in somatic symptoms | First visit of each patient at the Pain outpatient department of Hannover Medical School between 2019-02-28 and 2020-07-07
  Somatic symptoms assessed via the 15-item somatic scale (PHQ-15) from the German version of the Patient Health Questionnaire (PHQ-D). The score ranges from 0 (no somatic symptom burden) to 30 (maximal somatic symptom burden).
Difference in anxiety | First visit of each patient at the Pain outpatient department of Hannover Medical School between 2019-02-28 and 2020-07-07
  Anxiety assessed via the 7-item anxiety scale (GAD-7) from the German version of the Patient Health Questionnaire (PHQ-D). The score ranges from 0 (no anxiety) to 21 (maximal anxiety).
Difference in stress | First visit of each patient at the Pain outpatient department of Hannover Medical School between 2019-02-28 and 2020-07-07
  Stress assessed via the 10-item stress scale (PHQ-Stress) from the German version of the Patient Health Questionnaire (PHQ-D). The score ranges from 0 (no stress) to 20 (maximal stress).

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Manuel Sánchez, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Manuel J, Rudolph L, Beissner F, Neubert TA, Dusch M, Karst M. Traumatic Events, Posttraumatic Stress Disorder, and Central Sensitization in Chronic Pain Patients of a German University Outpatient Pain Clinic. Psychosom Med. 2023 May 1;85(4):351-357. doi: 10.1097/PSY.0000000000001181. Epub 2023 Feb 21. PMID 36825929